CLINICAL TRIAL: NCT00405769
Title: Alternative Lipid Lowering in Patients With Statin Intolerance: Use of Red Yeast Rice and Therapeutic Lifestyle Changes in a Randomized, Placebo-Controlled Trial
Brief Title: Lipid Lowering in Patients With Statin Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Hill Health System (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: FWA00005390
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Hyperlipidemia; Coronary Artery Disease
Keywords: statin intolerance; hyperlipidemia; lifestyle changes; red yeast rice
MeSH Terms: conditions — Hyperlipidemias; Coronary Artery Disease | interventions — red yeast rice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator): placebo control
  Interventions: Drug: placebo
- 2 (Active Comparator): red yeast rice
  Interventions: Drug: red yeast rice

INTERVENTIONS:
Drug: red yeast rice — 600 mg 3 caps bid
  Arms: 2
Drug: placebo — 3 caps bid
  Arms: 1

SUMMARY:
This study will attempt to further validate a clinical treatment plan to lower LDL values using non-prescription supplements combined with a lifestyle change and education program which could represent an alternative approach to improve compliance in group of people who are unable to take traditional medication to lower cholesterol.

DETAILED DESCRIPTION:
Up to 70 participants will be randomized into 2 groups. Each shall have similar total and LDL cholesterol values obtained prior to the study. Study Group 1 will participate in the Change of Heart Program (an intensive program to make therapeutic lifestyle changes) and take a placebo pill. Study Group 2 will also participate in Change of Heart. Group 2 will be provided an over the counter supplement consisting of red rice yeast 2.4-3.6 gms day)

Blood work consisting of a lipid panel, cardiac CRP, CPK, liver function panel and TSH will be obtained prior to study, and at 12 and 26 wks. Questionnaires will be administered regarding quality of life indexes, and ancillary symptom relief (i.e. degree of arthritis discomfort, generalized weakness) before, 12 and 26 weeks. After the Change of Heart program ends (12 weeks), participants will continue on study medication for a total of 6 months. A final questionnaire and final blood work will be obtained at 6 months, and at that point, medications can be discontinued.

ELIGIBILITY:
Inclusion criteria:

1. Baseline cholesterol - LDL more than 160 with one risk factor or LDL more than 130 with 2 or more risk factors for developing coronary artery disease (Smoker, age >40, male, Family history, diabetes, obesity) utilizing ATP III guidelines
2. Have had a statin prescribed by a doctor for high cholesterol, and have stopped medication because of side effects
3. Ability to exercise without physical restrictions
4. Ability to attend 12 week consecutive Change of Heart sessions
5. Not taking any cholesterol lowering medication for at least 1 month prior to initiation of trial. Not taking red yeast rice for at least 1 month prior.

Exclusion Criteria:

1. Any active cardiac problem including chest pain, angina, shortness of breath with minimal activity, or unstable angina/acute coronary syndrome within one year
2. Known intolerance to one of the study drugs
3. Physical limitation preventing aerobic exercise program, such as severe arthritis, peripheral vascular disease, congestive heart failure, or symptom limiting pulmonary disease
4. Uncontrolled hypertension (defined as SBP>180 mmHg or DBP > 100mmHg.
5. Heart attack, bypass surgery, or angioplasty/stent within 1 year of study
6. Triglyceride level more than 400 mg/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol levels at baseline, 12 weeks and 6 months in 2 groups in a lifestyle intervention program | 24 weeks

SECONDARY OUTCOMES:
HDL, TG, Total cholesterol, cardiac CRP, | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J Becker, MD, Principal Investigator — Chestnut Hill Health System
Locations (1):
- Chestnut Hill Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Becker DJ, Gordon RY, Halbert SC, French B, Morris PB, Rader DJ. Red yeast rice for dyslipidemia in statin-intolerant patients: a randomized trial. Ann Intern Med. 2009 Jun 16;150(12):830-9, W147-9. doi: 10.7326/0003-4819-150-12-200906160-00006. PMID 19528562